CLINICAL TRIAL: NCT03693027
Title: Evaluation of a Daily Oral Care Lozenge on Oral Health and Quality of Life in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Primal Therapies Inc. (Industry)
Collaborators: Benjamin Rose Institute on Aging (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2017-04
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Oral Health
Keywords: Older adults; microbiome; gum health; gingivitis; gum disease
MeSH Terms: conditions — Gingivitis; Gingival Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTx800 (Experimental): Qualified subjects will dissolve one oral lozenge (PTx800 lozenges) by mouth 3 times a day (after breakfast, lunch and dinner) throughout the 6 week study.
  Interventions: Dietary Supplement: PTx800 lozenges
- Placebo (Placebo Comparator): Qualified subjects will dissolve one oral lozenge (placebo control) by mouth 3 times a day (after breakfast, lunch and dinner) throughout the 6 week study.
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: PTx800 lozenges — PTX800 is a nutritional supplement containing generally recognized as safe designated active ingredients in a rapid melt oral lozenges.
  Arms: PTx800
Dietary Supplement: Placebo control — The placebo of PTX800 is a rapid melt oral lozenge without the active ingredients found in the PTX800 lozenges.
  Arms: Placebo

SUMMARY:
The assessment of a daily oral care lozenge (PTx800) will be compared to a placebo control in a cohort of older adults who visit adult senior centers and who also have mild to moderate gingivitis. The comparison of the pre-to post change in gum health and pathogen burdens will be measured over a 6 week period. In addition, the feasibility and acceptability of using the lozenges will be assessed in this older adult population.

DETAILED DESCRIPTION:
By 2030, 70 million Americans will be over the age of 65. Currently, 70% of older adults have periodontal disease, 20% have untreated tooth decay, and 1 in 4 older adults have lost some or all of their teeth. This poses a significant problem as mounting evidence demonstrates a link between oral disease and life-threatening diseases, including premature death. Gum disease is associated with systemic conditions such as cardiovascular disease, stroke, diabetes mellitus, chronic kidney disease, respiratory disorders, dementia and cancers. Moreover, numerous studies suggest that the number of teeth lost in adulthood is a predictor of premature death. Therefore, an individual's oral health and general health are tightly linked and good oral hygiene could be an easy means of preventing serious, life-threatening conditions in many older adults.

For many older adults, decreased manual dexterity, physical or mental impairment, income constraints, lack of dental insurance, all contribute to and exacerbate oral disease. A cost-effective, nontoxic and easy-to-take oral solution has been developed; PTx800 rapid dissolving lozenges. The investigators are evaluating PTx800 lozenge performance on gum health and ease of use in the older adult population who frequent community centers in the greater Cleveland, Ohio area. Efficacy assessment will be determined over the course of 6 weeks on participants with confirmed mild-to-moderate gingivitis. Endpoint measurements on gum health for PTx800 vs placebo control will be evaluated. Furthermore, the ease of use and receptivity to the PTx800 lozenges will be assessed in order to determine whether the PTx800 lozenges could be a viable candidate to supplement standard oral hygiene practices. A comparison in the change in oral health outcomes and dental pathogen burdens will be investigated in the 6-week study. As a part of the study design, a survey of this population will be conducted to understand perceptions, biases and habits as they relate to oral health, social and emotional well-being. The culmination of this work will impart a better understanding of, and facilitate appropriate actions to address, the oral health crisis in older adults. The ultimate goal of this study is to identify methods to improve the quality of life for this demographic.

ELIGIBILITY:
Inclusion Criteria:

* age range between 60 and 85 years,
* non-smokers or those who have stopped for 2 years or more,
* baseline gingival index (MGI score greater or equal to 1.75),
* score of 4 or lower on the Short Portable Mental Status Questionnaire (SPMSQ).

Exclusion Criteria:

* subjects on antibiotic within the previous 30 days,
* fixed or removable full dentures,
* advanced periodontitis,
* significant oral soft tissue pathology based on a visual examination (excluding gingivitis),
* gross dental caries,
* score of 5 or higher on the Short Portable Mental Status Questionnaire (SPMSQ).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-20 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of Bacterial Burden | Measured at baseline and at 6 weeks
  Oral swabs and oral mouth rinses will be taken from subjects. Bacterial burden and composition will be determined by live bacterial cultures and quantitative polymerase chain reaction.
Change from Baseline of Oral Health | Measured at baseline and at 6 weeks
  Oral gum health and dental assessments including modified gingival index will be determined by a licensed dental practitioner. The Modified Gingival Index (MGI) uses non-invasive/no probing methods. The scoring system rates mild and moderate inflammation where: 0 = no inflammation; 1 = mild inflammation or with slight changes in color and texture in a portion of gingival tissue; 2 = mild inflammation in all portions of the gingiva; 3 = moderate, bright surface inflammation, erythema, edema and/or hypertrophy of gingival marginal or papillary; 4 = severe inflammation: erythema, edema and/or marginal gingival hypertrophy or spontaneous bleeding, papillary, congestion or ulceration.

SECONDARY OUTCOMES:
Change from Baseline in oral health behaviors and habits | Measured at baseline and at 6 weeks
  Subjects are asked a comprehensive questionnaire regarding overall medical and dental health as well as oral and dental care habits and behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Emily Stein, Principal Investigator — Primal Therapies
Locations (1):
- Benjamin Rose Institute on Aging, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] LaMonte MJ, Genco RJ, Hovey KM, Wallace RB, Freudenheim JL, Michaud DS, Mai X, Tinker LF, Salazar CR, Andrews CA, Li W, Eaton CB, Martin LW, Wactawski-Wende J. History of Periodontitis Diagnosis and Edentulism as Predictors of Cardiovascular Disease, Stroke, and Mortality in Postmenopausal Women. J Am Heart Assoc. 2017 Mar 29;6(4):e004518. doi: 10.1161/JAHA.116.004518. PMID 28356279
- [Background] Abbayya K, Puthanakar NY, Naduwinmani S, Chidambar YS. Association between Periodontitis and Alzheimer's Disease. N Am J Med Sci. 2015 Jun;7(6):241-6. doi: 10.4103/1947-2714.159325. PMID 26199919
- [Background] Kaur S, White S, Bartold M. Periodontal Disease as a Risk Factor for Rheumatoid Arthritis: A Systematic Review. JBI Libr Syst Rev. 2012;10(42 Suppl):1-12. doi: 10.11124/jbisrir-2012-288. PMID 27820156
- [Background] Kamer AR, Dasanayake AP, Craig RG, Glodzik-Sobanska L, Bry M, de Leon MJ. Alzheimer's disease and peripheral infections: the possible contribution from periodontal infections, model and hypothesis. J Alzheimers Dis. 2008 May;13(4):437-49. doi: 10.3233/jad-2008-13408. PMID 18487851
- [Background] Maisonneuve P, Amar S, Lowenfels AB. Periodontal disease, edentulism, and pancreatic cancer: a meta-analysis. Ann Oncol. 2017 May 1;28(5):985-995. doi: 10.1093/annonc/mdx019. PMID 28453689
- [Background] Momen-Heravi F, Babic A, Tworoger SS, Zhang L, Wu K, Smith-Warner SA, Ogino S, Chan AT, Meyerhardt J, Giovannucci E, Fuchs C, Cho E, Michaud DS, Stampfer MJ, Yu YH, Kim D, Zhang X. Periodontal disease, tooth loss and colorectal cancer risk: Results from the Nurses' Health Study. Int J Cancer. 2017 Feb 1;140(3):646-652. doi: 10.1002/ijc.30486. Epub 2016 Nov 23. PMID 27778343
- [Background] Michaud DS, Joshipura K, Giovannucci E, Fuchs CS. A prospective study of periodontal disease and pancreatic cancer in US male health professionals. J Natl Cancer Inst. 2007 Jan 17;99(2):171-5. doi: 10.1093/jnci/djk021. PMID 17228001
- [Background] Fardini Y, Wang X, Temoin S, Nithianantham S, Lee D, Shoham M, Han YW. Fusobacterium nucleatum adhesin FadA binds vascular endothelial cadherin and alters endothelial integrity. Mol Microbiol. 2011 Dec;82(6):1468-80. doi: 10.1111/j.1365-2958.2011.07905.x. Epub 2011 Nov 15. PMID 22040113
- [Background] Lamster IB. Oral health care services for older adults: a looming crisis. Am J Public Health. 2004 May;94(5):699-702. doi: 10.2105/ajph.94.5.699. No abstract available. PMID 15117682
- [Background] McClearn GE, Svartengren M, Pedersen NL, Heller DA, Plomin R. Genetic and environmental influences on pulmonary function in aging Swedish twins. J Gerontol. 1994 Nov;49(6):264-8. doi: 10.1093/geronj/49.6.m264. PMID 7963289
- [Background] Lee KH, Wu B, Plassman BL. Cognitive function and oral health-related quality of life in older adults. J Am Geriatr Soc. 2013 Sep;61(9):1602-7. doi: 10.1111/jgs.12402. Epub 2013 Aug 26. PMID 24028360
- [Background] Park H, Suk SH, Cheong JS, Lee HS, Chang H, Do SY, Kang JS. Tooth loss may predict poor cognitive function in community-dwelling adults without dementia or stroke: the PRESENT project. J Korean Med Sci. 2013 Oct;28(10):1518-21. doi: 10.3346/jkms.2013.28.10.1518. Epub 2013 Sep 25. PMID 24133359
- [Background] Del Brutto OH, Gardener H, Del Brutto VJ, Maestre GE, Zambrano M, Montenegro JE, Wright CB. Edentulism associates with worse cognitive performance in community-dwelling elders in rural Ecuador: results of the Atahualpa project. J Community Health. 2014 Dec;39(6):1097-100. doi: 10.1007/s10900-014-9857-3. PMID 24627152
- [Background] Lee KH, Plassman BL, Pan W, Wu B. Mediation Effect of Oral Hygiene on the Relationship Between Cognitive Function and Oral Health in Older Adults. J Gerontol Nurs. 2016 May 1;42(5):30-7. doi: 10.3928/00989134-20151218-03. Epub 2015 Dec 29. PMID 26716459
- [Background] Joshy G, Arora M, Korda RJ, Chalmers J, Banks E. Is poor oral health a risk marker for incident cardiovascular disease hospitalisation and all-cause mortality? Findings from 172 630 participants from the prospective 45 and Up Study. BMJ Open. 2016 Aug 30;6(8):e012386. doi: 10.1136/bmjopen-2016-012386. PMID 27577588
- [Background] Ruokonen H, Nylund K, Furuholm J, Meurman JH, Sorsa T, Kotaniemi K, Ortiz F, Heikkinen AM. Oral Health and Mortality in Patients With Chronic Kidney Disease. J Periodontol. 2017 Jan;88(1):26-33. doi: 10.1902/jop.2016.160215. Epub 2016 Aug 13. PMID 27523518
- [Background] Beukers NG, van der Heijden GJ, van Wijk AJ, Loos BG. Periodontitis is an independent risk indicator for atherosclerotic cardiovascular diseases among 60 174 participants in a large dental school in the Netherlands. J Epidemiol Community Health. 2017 Jan;71(1):37-42. doi: 10.1136/jech-2015-206745. Epub 2016 Aug 8. PMID 27502782
- [Background] Friedman PK, Lamster IB. Tooth loss as a predictor of shortened longevity: exploring the hypothesis. Periodontol 2000. 2016 Oct;72(1):142-52. doi: 10.1111/prd.12128. PMID 27501497
- [Background] Padilha DM, Hilgert JB, Hugo FN, Bos AJ, Ferrucci L. Number of teeth and mortality risk in the Baltimore Longitudinal Study of Aging. J Gerontol A Biol Sci Med Sci. 2008 Jul;63(7):739-44. doi: 10.1093/gerona/63.7.739. PMID 18693229
- [Background] American Dental Association Health Policy Institute. HPI: unmet dental needs falling for children, rising for low-income adults, seniors. ADA News. Sept 27, 2016.
- [Background] US Department of Health and Human Services. Oral Health in America: A Report of the Surgeon General- Executive Summary. Rockville, MD: US Department of Health and Human Services, National Institute of Dental and Craniofacial Research, National Institutes of Health, 2000.
- [Background] CDC report 2004: https://www.cdc.gov/aging/pdf/ state_of_aging_and_health_in_america_2004.pdf
- [Background] Shay K. Infectious complications of dental and periodontal diseases in the elderly population. Clin Infect Dis. 2002 May 1;34(9):1215-23. doi: 10.1086/339865. Epub 2002 Apr 2. PMID 11941548
- [Background] Persson RE, Persson GR. The elderly at risk for periodontitis and systemic diseases. Dent Clin North Am. 2005 Apr;49(2):279-92. doi: 10.1016/j.cden.2004.10.006. PMID 15755405
- [Background] Komiya K, Rubin BK, Kadota JI, Mukae H, Akaba T, Moro H, Aoki N, Tsukada H, Noguchi S, Shime N, Takahashi O, Kohno S. Prognostic implications of aspiration pneumonia in patients with community acquired pneumonia: A systematic review with meta-analysis. Sci Rep. 2016 Dec 7;6:38097. doi: 10.1038/srep38097. PMID 27924871
- [Background] Marsh PD, Zaura E. Dental biofilm: ecological interactions in health and disease. J Clin Periodontol. 2017 Mar;44 Suppl 18:S12-S22. doi: 10.1111/jcpe.12679. PMID 28266111
- [Background] Gross EL, Beall CJ, Kutsch SR, Firestone ND, Leys EJ, Griffen AL. Beyond Streptococcus mutans: dental caries onset linked to multiple species by 16S rRNA community analysis. PLoS One. 2012;7(10):e47722. doi: 10.1371/journal.pone.0047722. Epub 2012 Oct 16. PMID 23091642
- [Background] Peterson SN, Snesrud E, Liu J, Ong AC, Kilian M, Schork NJ, Bretz W. The dental plaque microbiome in health and disease. PLoS One. 2013;8(3):e58487. doi: 10.1371/journal.pone.0058487. Epub 2013 Mar 8. PMID 23520516
- [Background] Hajishengallis G, Liang S, Payne MA, Hashim A, Jotwani R, Eskan MA, McIntosh ML, Alsam A, Kirkwood KL, Lambris JD, Darveau RP, Curtis MA. Low-abundance biofilm species orchestrates inflammatory periodontal disease through the commensal microbiota and complement. Cell Host Microbe. 2011 Nov 17;10(5):497-506. doi: 10.1016/j.chom.2011.10.006. Epub 2011 Oct 27. PMID 22036469
- [Background] Hajishengallis G, Lamont RJ. Beyond the red complex and into more complexity: the polymicrobial synergy and dysbiosis (PSD) model of periodontal disease etiology. Mol Oral Microbiol. 2012 Dec;27(6):409-19. doi: 10.1111/j.2041-1014.2012.00663.x. Epub 2012 Sep 3. PMID 23134607
- [Background] CDC report 2008 https://www2c.cdc.gov/podcasts/media/pdf/ HealthyAging_OralHealth.pdf
- [Background] Fox PC and Eversole LR. Diseases of the salivary glands. In: Silverman S, Eversole LR, Truelove EL, eds. Essentials of Oral Medicine. Ontario, Canada: BC Decker; 2002:260-276
- [Background] From Medicare website: (https://www.medicare.gov/coverage/dentalservices. html).